



A Phase 2 Multiple Dose Study to Evaluate the Efficacy and Safety of PUL-042 Inhalation Solution in Reducing the Infection Rate and Progression to COVID-19 in Adults Exposed to SARS-CoV-2

Protocol Number: PUL-042-501

Protocol Version: 1.60

Protocol Date: 29 January 2021

# STATISTICAL ANALYSIS PLAN

Version 1.0




# A Phase 2 Multiple Dose Study to Evaluate the Efficacy and Safety of PUL-042 Inhalation Solution in Reducing the Infection Rate and Progression to COVID-19 in Adults Exposed to SARS-CoV-2

# STATISTICAL ANALYSIS PLAN

Version 1.0

**Author:** Yuhui Qiu

Principal Biostatistician, CTI

**CTI Biostatistics** 

**Reviewer:** David McCollum

Director, Global Biostatistics, CTI

**Sponsor Approval:** Colin Broom

Chief Executive Officer

Pulmotect, Inc.




# **Table of Contents**

| LIS | ST OF ABBREVIATIONS | 5 |
|---|---|---|
| 1. | INTRODUCTION | 6 |
| 2. | OBJECTIVES AND ENDPOINTS | |
| | 2.1 Objectives | 6 |
| 4 | 2.1.1 Primary Objective | |
| | 2.1.2 Secondary Objectives | |
| 2 | 2.2 Endpoints | |
| | 2.2.1 Primary Efficacy Endpoint | |
| | 2.2.2 Secondary Efficacy Endpoints | |
| | 2.2.3 Safety and Tolerability Endpoints | 7 |
| 3. | INVESTIGATIONAL PLAN | 7 |
| | 3.1 STUDY DESIGN | 7 |
| | 3.2 Treatment | |
| | 3.2.1 Randomization Scheme and Treatment Arm Assignment | |
| | 3.2.2 Blinding | |
| | 3.2.3 Dosing Schedule | 8 |
| | 3.2.4 Subject Compliance | 8 |
| 4. | CENERAL CONSIDERATIONS FOR DATA ANALYSIS | 8 |
| 5. | | |
| 4 | 5.1 DISPOSITION OF SUBJECTS | .10 |
| 4 | 5.2 PROTOCOL DEVIATIONS | .11 |
| 4 | 5.3 DEMOGRAPHIC CHARACTERISTICS | |
| | 5.4 Baseline Characteristics | |
| | 5.6 CONCOMITANT MEDICATIONS AND PROCEDURES | .11 |
| 6. | EFFICACY ANALYSES | .12 |
| ( | 5.1 PRIMARY EFFICACY ENDPOINT AND ANALYSIS | .12 |
| 6 | 5.2 SECONDARY EFFICACY ENDPOINTS AND ANALYSES | .13 |
| | Incidence of SARS-CoV-2 infection through Day 29 | .13 |
| | Incidence of SARS-CoV-2 infection through Day 15 | .13 |
| | Severity of COVID-19 through Day 15 | |
| | Ordinal Scale through Day 29 | |
| | Symptom Score | |
| | Subjects requiring ICU admission | edule 8 npliance 8 IDERATIONS FOR DATA ANALYSIS 8 Y ASSURANCE 9 S. 9 WINDOWS 10 DROPOUTS OR MISSING DATA 10 MPARISONS 10 TIONS AND TRANSFORMATIONS 10 IS 10 IF SUBJECTS 10 VIATIONS 11 C CHARACTERISTICS 11 TORY 11 I MEDICATIONS AND PROCEDURES 11 LYSES 12 CACY ENDPOINT AND ANALYSIS 12 FFICACY ENDPOINTS AND ANALYSIS 12 FFICACY ENDPOINTS AND ANALYSIS 13 CoV-2 infection through Day 29 13 CoV-2 infection through Day 15 13 19 through Day 15 13 19 through Day 15 13 19 through Day 29 14 CU admission 14 |
| | Number of ICU Days | |
| | Subjects requiring mechanical ventilation | .13 |



| Λ | Number of days on mechanical ventilation | |
|------|------------------------------------------------|----|
| | Nortality Rate through Day 29 | |
| 6.3 | SUBGROUP ANALYSES | 16 |
| 7. S | SAFETY AND TOLERABILITY ANALYSIS | 16 |
| 7.1 | EXTENT OF EXPOSURE AND COMPLIANCE | 16 |
| 7.2 | ADVERSE EVENTS | 17 |
| 7. | 7.2.1 Treatment-emergent Adverse Events | |
| 7. | 7.2.2 Adverse Event Severity | 17 |
| 7. | 7.2.3 Adverse Event Relationship to Study Drug | 17 |
| 7. | 7.2.4 Serious Adverse Events | |
| 7. | 7.2.5 Adverse Event Summaries | |
| 7.3 | PULMONARY FUNCTION TESTING | 19 |
| 7.4 | VITAL SIGNS | |
| 7.5 | OTHER SAFETY MEASURES | 19 |
| 8. I | NTERIM ANALYSES | 20 |
| 9. S | SAMPLE SIZE AND POWER CALCULATIONS | 20 |
| 10. | REFERENCES | 20 |
| 11. | APPENDIX | 21 |
| 11.1 | APPENDIX A: SCHEDULE OF EVENTS | 21 |



# LIST OF ABBREVIATIONS

| Abbreviation | Definition |
|---|---|
| ADL | Activities of Daily Living |
| AE | Adverse event |
| ATC | Anatomical, Therapeutic, and Chemical |
| BMI | Body mass index |
| CI | Confidence interval |
| СМН | Cochran-Mantel-Haenszel |
| CTCAE | Common Terminology Criteria for Adverse Events |
| COVID-19 | Coronavirus Disease 2019 caused by the SARS-CoV-2 virus |
| DSMB | Data and Safety Monitoring Board |
| eCRF | Electronic Case Report Form |
| FEV1 | forced expiratory volume in 1 second |
| ICU | Intensive care unit |
| ITT | Intention to Treat |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mITT | Modified Intention to Treat |
| ODN | ODN M362 |
| Pam2 | Pam2CSK4 |
| PI | Principal Investigator |
| PT | Preferred term |
| PUL-042 | drug product consisting of a 4:1 molar ratio of Pam2:ODN;<br>Inhalation Solution |
| SAE | Serious adverse event |
| SAF | Safety |
| SAP | Statistical analysis plan |
| SARS-CoV-2 | Coronavirus causing COVID-19 |
| SOC | System organ class |
| TEAE | Treatment-emergent adverse event |
| WHO | World Health Organization |




#### 1. INTRODUCTION

This statistical analysis plan (SAP) is based on the Protocol # PUL-042-501 Version 1.60, dated 19 January 2021, and titled "A Phase 2 Multiple Dose Study to Evaluate the Efficacy and Safety of PUL-042 Inhalation Solution in Reducing the Infection Rate and Progression to COVID-19 in Adults Exposed to SARS-CoV-2." See the study protocol for full details.

This document details the statistical methods planned to perform the analysis for Data Safety Monitoring Board (DSMB), as well as the final analysis of the study.

## 2. OBJECTIVES AND ENDPOINTS

# 2.1 Objectives

# 2.1.1 Primary Objective

To determine the efficacy of PUL-042 Inhalation Solution in the prevention of viral infection with SARS-CoV-2 and progression to COVID-19 in subjects: 1) who have repeated exposure to individuals with SARS-CoV-2 infection, and 2) are asymptomatic at enrollment.

# 2.1.2 Secondary Objectives

- To determine the difference in incidence of SARS-CoV-2 infection 28 days from the start of experimental therapy in subjects who test negative for SARS-CoV-2 at the pre-treatment visit
- To determine the difference in incidence of SARS-CoV-2 infection 14 days from the start of experimental therapy in subjects who test negative for SARS-CoV-2 at the pre-treatment visit
- To compare the severity of COVID-19 within 14 days from the start of experimental therapy
- To compare the severity of COVID-19 within 28 days from the start of experimental therapy
- To assess the requirement for ICU admission within 28 days from the start of experimental therapy
- To assess the requirement for mechanical ventilation within 28 days from the start of experimental therapy
- To assess mortality within 28 days from the start of experimental therapy
- To determine the tolerability of PUL-042 Inhalation Solution in this population

# 2.2 Endpoints

# 2.2.1 Primary Efficacy Endpoint

The primary endpoint is the severity of COVID-19 as measured by the maximum difference from the baseline value in the Ordinal Scale for Clinical Improvement within 28 days from the start of experimental therapy.




# 2.2.2 Secondary Efficacy Endpoints

The secondary efficacy endpoints include the following:

- Incidence of SARS-CoV-2 infection 28 days from the start of experimental therapy in subjects who test negative for SARS-CoV-2 at the pre-treatment visit
- Incidence of SARS-CoV-2 infection 14 days from the start of experimental therapy in subjects who test negative for SARS-CoV-2 at the pre-treatment visit
- Severity of COVID-19 as measured by the maximum difference from the baseline value in the Ordinal Scale for Clinical Improvement within 14 days from the start of experimental therapy.
- Ordinal Scale for Clinical Improvement within 28 days from the start of experimental therapy
- SARS-Cov-2 Symptom Score during the study
- Proportion of subjects requiring ICU admission from Day 1 to Day 29
- Number of ICU Days from Day 1 to Day 29
- Proportion of subjects requiring mechanical ventilation from Day 1 to Day 29
- Number of days on mechanical ventilation from Day 1 to Day 29
- All-cause mortality rate through Day 29

# 2.2.3 Safety and Tolerability Endpoints

- Reduction in forced expiratory volume in 1 second (FEV1) from Pre-dose to Post-dose
- Treatment-emergent serious adverse events (SAEs) through Day 29
- Treatment-emergent adverse events (TEAEs) and severity through Day 29
- Vital signs

#### 3. INVESTIGATIONAL PLAN

### 3.1 Study Design

This will be a double-blind trial. A total of approximately 200 subjects randomized 1:1 (PUL-042 Inhalation Solution: placebo) will be enrolled in the trial.

Doses will be administered via nebulization with a PARI Sprint nebulizer. All subjects will receive up to 4 doses of PUL-042 Inhalation Solution or placebo over 10 days (Days 1, 3, 6, and 10).

Subjects will participate for approximately 28 days. See Appendix A for the Schedule of Events.

An overview of the study design is presented below:






#### 3.2 Treatment

# 3.2.1 Randomization Scheme and Treatment Arm Assignment

Subjects will be randomly assigned to receive PUL-042 Inhalation Solution or placebo in a 1:1 ratio. A central randomization system, the Medication Assignment Center (MAC; CTI Clinical Trial and Consulting Services), will be used for this study.

# 3.2.2 Blinding

The sponsor, subjects, Principal Investigator (PI), and site study staff (except for the unblinded study drug personnel) will not know the treatment (PUL-042 vs. placebo) a subject receives. The CRO staff dealing with blinded site study staff and the study statistician will also be blinded. The statistician who generates the production randomization code, MAC Operators who perform the randomization and the unblinded study team will be unblinded to the treatment a subject receives.

All doses of study drug (i.e., both Active and Placebo) will be prepared at the site, so the site Pharmacists will also be unblinded.

# 3.2.3 Dosing Schedule

The dose level of PUL-042 Inhalation Solution in this study will be 20.3  $\mu$ g Pam2 : 29.8  $\mu$ g ODN/mL (50  $\mu$ g PUL-042). A total of up to 4 doses will be administered over a 10-day period for a total dose of 81.2  $\mu$ g Pam2 : 119.2  $\mu$ g ODN.

Doses of PUL-042 or placebo will be prepared by an unblinded pharmacist and administered to the subject within 4 hours of preparation.

Doses will be administered via nebulization to deliver 4 mL using a PARI Sprint nebulizer equipped with a filter valve to prevent aerosol generation. The nebulizer will be operated until all drug is delivered.

# 3.2.4 Subject Compliance

Any material deviation from study procedures (identified by site personnel or monitor) will be documented. Major subject-level deviations will be captured on the protocol deviation form. A list of protocol deviations will be compiled and reviewed by the PI and Sponsor to identify major and minor deviations periodically using the criteria specified in the Protocol, Section 14.5.

# 4. GENERAL CONSIDERATIONS FOR DATA ANALYSIS

Unless otherwise specified, continuous variables will be summarized using descriptive statistics (n, mean, standard deviation, median, minimum, and maximum). Categorical variables will be summarized showing the number and percentage of subjects within each category.




Summary results will be provided for each treatment group. All tabulations will be based on pooled data across centers.

Unscheduled visits will be excluded from the summaries but will be included in the data listings.

All statistical tests will be two-sided and tested at the 10% level of significance.

Analyses will be performed using SAS for Windows statistical software, version 9.4 or higher (SAS, Cary, NC), except where other software may be deemed more appropriate.

CTI will perform all efficacy and safety analyses described in this SAP.

Subject data will be listed, sorted by treatment group and subject number. When applicable, listings will be additionally sorted by visit and assessment date/time.

# 4.1 Data Quality Assurance

Once all the source verification is complete, all queries are resolved, and the database has been updated appropriately, the database will be locked and made available to CTI Biostatistics for final analysis.

Data may be pulled by CTI Biostatistics for DSMB analysis at a time when source verification and query resolution is ongoing.

All SAS programs used to create analysis data sets, tables, and listings are double programmed. The SAS outputs will be compared and the programs will be updated until the outputs match.

# 4.2 Analysis Sets

The following three analysis sets will be defined for this study:

# Intent to Treat (ITT) Set

The ITT set is defined as all randomized subjects who receive at least one dose of experimental treatment (i.e., PUL-042 or Placebo). Randomized subjects are to be symptoms free and not known to be SARS-CoV-2 positive at baseline. The primary analysis of the efficacy endpoints will be carried out using the ITT set based on the randomized treatment, except for the first two secondary efficacy endpoints listed in Section 2.2.2.

#### Modified Intent to Treat (mITT) Set

The mITT set will include all randomized subjects who receive at least one dose of experimental treatment (i.e., PUL-042 or Placebo) and are negative for SARS-CoV-2 infection at the time of administration of the first dose.

The mITT set will be used for the analyses of the first two secondary efficacy endpoints listed in Section 2.2.2.

## Safety (SAF) Set

The SAF set is also defined as all randomized subjects who receive at least one dose of experimental treatment (i.e., PUL-042 or Placebo), but subjects are categorized based on the treatment actually received rather than as randomized. All safety and tolerability analyses will be carried out using the SAF set. If, as is expected, the Safety analysis set is redundant (i.e., is identical to the ITT analysis set), the ITT set will be used for the assessments of safety and tolerability.




#### 4.3 Assessment Windows

Data will be summarized by nominal study visit recorded in the database.

# 4.4 Handling of Dropouts or Missing Data

Except for the time to event endpoint (Table 1), partial end dates of prior and concomitant medications (Section 5.6), and partial onset dates of AEs (Section 7.2.1), all other missing data will be treated as missing and no method for imputation is planned.

Missing data on the time to event endpoint will have events coded as right censored per the following table:

**Table 1 Missing Data Coding for Time to Event Data Analysis** 

| Endpoint | Right Censoring |
|---|---|
| Subject Survival | Subjects who are still alive as of the last known follow-up will be right censored as of the date of last subject contact when the subject was known to be alive. |

# 4.5 Multiple Comparisons

Because of the exploratory nature of this study, there will be no adjustment for multiple comparisons.

#### 4.6 Data Derivations and Transformations

The following derivations will be used in this study:

Study Day (Note: There is no day 0 in this study):

- Date of assessment date of 1<sup>st</sup> Study Drug administration + 1 for assessments done on or after date of 1<sup>st</sup> Study Drug administration
- Date of assessment date of 1<sup>st</sup> Study Drug administration for assessments done before date of 1<sup>st</sup> Study Drug administration

Baseline Observation: the last non-missing value prior to 1<sup>st</sup> Study Drug administration.

# **Duration**:

- Duration in days = end date start date + 1
- Duration in minutes = end time in minutes start time in minutes

# 5. STUDY SUBJECTS

# 5.1 Disposition of Subjects

A table of frequency counts and percentages of all subjects who are randomized, and in each analysis set will be provided. Subject disposition including study completion status and reasons for early termination will be tabulated by treatment group and overall. A by subject listing will be provided.




#### **5.2** Protocol Deviations

Distribution of the types of protocol deviations and the number of subjects that deviate from the protocol will be tabulated for the treatment groups in the ITT set. Protocol deviations will also be tabulated by severity (e.g., minor or major) if appropriate. A listing of all protocol deviations will be provided.

# **5.3** Demographic Characteristics

Descriptive statistics will be used to summarize the demographic characteristics (age, gender, race, ethnicity, height, weight, and Body Mass Index [BMI]) for the ITT set. A by subject listing will be provided.

#### 5.4 Baseline Characteristics

Baseline characteristics of ITT subjects including SARS-CoV-2 exposure and spirometry results at Screening will be listed and tabulated.

# 5.5 Medical History

All medical conditions and surgical procedures will be classified by system organ class (SOC) and preferred term (PT) using the Medical Dictionary for Regulatory Activities (MedDRA). The number and percent of subjects with each medical condition and surgical procedure will be presented for each SOC and PT for the ITT set.

#### 5.6 Concomitant Medications and Procedures

All concomitant medications collected will be coded using the World Health Organization (WHO) Drug Dictionary. The number and percent of ITT subjects using concomitant medications will be tabulated by Anatomical, Therapeutic, and Chemical (ATC) level 2 and by preferred name. If the ATC level 2 is missing, the higher ATC level term will be used in the medication summary table and data listing.

A listing of all medications will be provided. The listing will include flags for prior medications.

Prior medications are defined as medications that ended prior to the date of first Study Drug administration. Concomitant medications are defined as medications that started at any time but ended on or after the date of first Study Drug administration, including those that are ongoing at study completion. In the case of a partial end date/time, in order to determine whether a medication is prior or concomitant, the following conservative imputation rule will be used: the unknown portions of a medication end date will be imputed to the latest possible. The imputed medication end date will then be compared with the date of first Study Drug administration to determine if the medication is prior or concomitant.

Note the imputed end date will only be used to determine whether a medication is prior or concomitant. The actual date reported on the electronic case report forms (eCRFs) will be presented in the listing.

Concomitant procedures will be collected via free text in the eCRF. These data will be presented in a listing.




#### 6. EFFICACY ANALYSES

Data on all efficacy endpoints will be listed and tabulated as appropriate.

# 6.1 Primary Efficacy Endpoint and Analysis

The primary efficacy analysis will be carried out on the ITT set.

The primary efficacy variable is the severity of COVID-19 as measured by the maximum difference from the baseline value in the Ordinal Scale for Clinical Improvement within 28 days from the start of experimental therapy. Randomized subjects are to be symptoms free and not known to be SARS-CoV-2 positive at baseline.

The Ordinal Scale for Clinical Improvement is a 9-point scale that measures disease severity at a given point in time. Notably, a score of 0 indicates that an individual is infection-free. The difference in scores obtained at different times provides a quantitative assessment of the incidence of infection and change in disease severity over that time interval.

The Ordinal Scale for Clinical Improvement to be used in this study is derived from a draft scale proposed by the World Health Organization<sup>[1]</sup> for clinical improvement as presented below:

Table 2 Ordinal Scale for Clinical Improvement (Derived from draft WHO scale)<sup>[1]</sup>

| Descriptor | Score |
|---|---|
| No clinical or virological evidence of infection | 0 |
| Infected but no limitation of activities | 1 |
| Limitation of activities | 2 |
| Hospitalized not requiring oxygen therapy (SpO2 > 93% on room air) | 3 |
| Oxygen by mask or nasal prongs | 4 |
| Non-invasive ventilation or high-flow oxygen | 5 |
| Intubation and mechanical ventilation | 6 |
| Ventilation + additional organ support- pressors, RRT, ECMO | 7 |
| Death | 8 |

The null hypothesis is that there is no difference in mean maximum change in Ordinal scale from baseline through Day 29 between randomized treatment groups; H<sub>0</sub>:  $\Delta_t$  -  $\Delta_c$  = 0. The alternative hypothesis is that the mean maximum change in Ordinal scale from baseline through Day 29 are different between the treatment groups; H<sub>1</sub>:  $\Delta_t$  -  $\Delta_c \neq 0$ .

The change in severity of COVID-19 between the placebo- and actively-treated groups will be compared using an analysis of covariance (ANCOVA) model, including the maximum change in




Ordinal scale from baseline through Day 29 as a dependent variable, treatment group as a fixed effect, and baseline characteristics such as age as a covariate.

From this model, the least-squares (LS) means and 90% CIs for each treatment group, the treatment difference in the LS means, the 90% CI for the difference, and the associated p-value will be presented.

If the data cannot support ANCOVA model assumption, a sensitivity analysis will be performed using proportional-odds cumulative logit model. The cumulative logits model will compare lower ordinal scales to higher ones, or equivalently, more favorable outcomes to less favorable ones. The model may be adjusted for baseline characteristics such as age, if appropriate. The estimated odds ratio and 95% CI will be presented.

The proportional odds assumption will be tested using a score test at the two-sided alpha level of 0.05. In the event that the proportional odds assumption is not satisfied, given the anti-conservative nature of the score test, the proportional odds model will still be used for the analysis, and the results will be presented along with the score test p-value to help put these results in context. If the proportion odds assumption is rejected or if the proportional odds model fails to converge, an alternative analysis using Cochran-Mantel-Haenszel (CMH) test will be performed to evaluate the association between the treatment groups and the maximum change in ordinal scale from baseline. The p-value for CMH row mean scores statistic will be reported.

# 6.2 Secondary Efficacy Endpoints and Analyses

# **Incidence of SARS-CoV-2 infection through Day 29**

The analysis of the proportion of subjects who had a positive result from the SARS-CoV-2 test within 28 days from the first dose of study drug will be performed using the mITT set.

The null hypothesis is that there is no difference in proportions of subjects with SARS-CoV-2 infection through Day 29 between randomized treatment groups;  $H_0$ :  $\pi_t$  -  $\pi_c$  = 0. The alternative hypothesis is that the proportions of subjects with SARS-CoV-2 infection through Day 29 are different between the treatment groups;  $H_1$ :  $\pi_t$  -  $\pi_c \neq 0$ .

The proportion of mITT subjects with SARS-CoV-2 infection within each treatment group will be presented along with a two-sided exact (Clopper-Pearson) 90% confidence interval (CI).

The observed difference in the proportion of subjects with SARS-CoV-2 infection between treatment groups along with the exact unconditional 90% CI for risk difference will be calculated. The null hypothesis will be tested using Fisher's exact method and the p-value will be reported.

#### **Incidence of SARS-CoV-2 infection through Day 15**

The analysis of the proportion of mITT subjects who had a positive result from SARS-CoV-2 test within 14 days from the first dose of study drug will be performed using the method described above for the analysis of incidence of SARS-CoV-2 infection through Day 29.

## **Severity of COVID-19 through Day 15**

The change in severity of COVID-19 from baseline through Day 15 between the treatment groups will be compared using an ANCOVA model, including the maximum change in Ordinal scale from baseline through Day 15 as a dependent variable, treatment group as a fixed effect, and baseline




characteristics such as age as a covariate.

From this model, the least-squares (LS) means and 90% CIs for each treatment group, the treatment difference in the LS means, the 90% CI for the difference, and the associated p-value will be presented.

If the data cannot support ANCOVA model assumption, a sensitivity analysis will be performed using proportional-odds cumulative logit model as described above for the primary efficacy endpoint analysis.

# **Ordinal Scale through Day 29**

The absolute value and change from baseline in the Ordinal scale from Day 1 through Day 29 will be summarized by treatment group and visit using descriptive statistics.

The number and percentages of subjects in each severity category of the 9-point Ordinal Scale will be presented by visit and treatment group.

Graphical illustrations of the Ordinal Scales through Day 29 will be presented using stacked bar chart for each treatment group. The X axis representing time points and Y axis representing the cumulative number of subjects for each Ordinal Scale. Each bar is divided into a number of subbars stacked end to end corresponding to different Ordinal Scales.

The changes in Ordinal Scales through Day 29 will be examined using box and whisker plots for each treatment group. The X axis representing the post-baseline time points and the Y axis representing the change from baseline in Ordinal Scales at each post-baseline visit.

## **Symptom Score**

The symptoms due to SARS-CoV-2 infection will be assessed and the symptom scores (Cough (0-3), Shortness of breath or difficulty breathing (0-3), Muscle aches or fatigue (0-3), Fever (0-4)) will be recorded in the eCRF.

The respiratory symptom score will be calculated by summing the symptom scores from Cough and Shortness of breath or difficulty breathing. The total symptom score will be calculated by summing all symptom scores.

The scores from each symptom together with calculated respiratory symptom scores and total symptom scores will be summarized by presenting the number and percentage of ITT subjects for each category by visit and treatment group.

Each symptom score (Cough, Shortness of breath or difficulty breathing, Fatigue, Fever, Respiratory, Total) from each post-baseline timepoint will be compared between treatment groups using non-parametric Wilcoxon Rank Sum test at 2-sided alpha level of 0.1. The p-value will be presented at each post-baseline visit.

A radar plot will be created by presenting each symptom score in group mean at each time point by treatment group.

# **Subjects requiring ICU admission**

Subject data pertaining to ICU admission will be recorded in the database.

The proportion of ITT subjects who are admitted to the ICU from Day 1 to Day 29 within each




treatment group will be presented along with a two-sided exact (Clopper-Pearson) 90% confidence interval (CI).

The observed difference in the proportion of subjects requiring ICU admission between treatment groups along with the exact unconditional 90% CI for risk difference will be calculated. The null hypothesis will be tested using Fisher's exact method and the p-value will be reported.

Subjects who have died without ICU admission during the study will be counted as requiring ICU admission for the analysis.

### **Number of ICU Days**

The number of ICU days from Day 1 to Day 29 will be calculated based on the ICU admission and discharge dates recorded in the eCRF. The calculated number of ICU days will be compared between treatment groups using 2-sided Student's t-test. The 90% CI and p-value will be presented.

If the Student's t-test normality assumption is found to be clearly violated, a sensitivity analysis will be performed using a non-parametric Wilcoxon rank-sum test. The p-value from the test will be presented.

Subjects who died will be assigned as hospitalized in the ICU for the number of days remaining from the day of death to Day 29 for the analysis. Subjects who are alive and never admitted into the ICU will be included in the analysis with a value of zero ICU days.

Subjects who were at ICU at study completion will be assigned an ICU end date equal to the date of completion for the purpose of deriving number of ICU days.

## **Subjects requiring mechanical ventilation**

Subject data pertaining to mechanical ventilation use will be recorded in the database.

The proportion of ITT subjects who were on mechanical ventilation from Day 1 to Day 29 within each treatment group will be analyzed and compared using the method described above for the analysis of subjects requiring ICU admission.

Subjects who have died without mechanical ventilation during the study will be counted as requiring mechanical ventilation for the analysis.

#### Number of days on mechanical ventilation

The number of days on mechanical ventilation from Day 1 through Day 29 will be calculated based on the start/stop dates of mechanical ventilation recorded in the eCRF. Number of days on mechanical ventilation will be compared between treatment groups using 2-sided Student's t-test. The 90% CI and p-value will be presented.

If the Student's t-test normality assumption is found to be clearly violated, a sensitivity analysis will be performed using a non-parametric Wilcoxon rank-sum test. The p-value from the test will be presented.

Subjects who died will be assigned as being on mechanical ventilation for the number of days remaining to Day 29 for the analysis. Subjects who had mechanical ventilation ongoing at study completion will be assigned a mechanical ventilation end date equal to the date of study completion for the purpose of deriving duration of mechanical ventilation. Subjects who are alive and never




placed on mechanical ventilation will be included in the analysis with a value of zero days on mechanical ventilation.

### **Mortality Rate through Day 29**

Subject status (Alive/Death) will be recorded in the database. If the vital status of the subject is missing at the end of the study, then the subject will be excluded from the binomial analysis for the mortality rate. The subject will be included in the Kaplan-Meier (KM) analysis with right censoring at the date the subject was last known to be alive.

The mortality rate (proportion of ITT subjects who die) through Day 29 within each treatment group will be presented along with a two-sided exact (Clopper-Pearson) 90% confidence interval (CI).

The observed difference in the mortality rate between treatment groups along with the exact unconditional 90% CI for risk difference will be calculated. The null hypothesis will be tested using Fisher's exact method and the p-value will be reported.

If deemed appropriate, an alternative analysis will be performed in which the survival rates will be estimated using the KM method. The KM estimates along with 90% CIs and survival curves will be provided. Based on the KM estimates, the survival probabilities and associated 90% CIs on Days 15 and 29 will be reported; in addition, the 25%, 50% (median), and 75% percentiles of the survival time with associated 90% CIs will be provided, as data permit. The survival rates between treatment groups will be compared using Log-rank test and the p-value from Log-rank test will be presented.

## 6.3 Subgroup Analyses

Exploratory subgroup analyses of the primary efficacy endpoint by baseline characteristics, e.g. age group and gender, will be performed using the analysis method described in Section 6.1, if appropriate.

Additional analyses may be performed to gain a better understanding but would not replace analyses planned for primary and secondary efficacy endpoints.

#### 7. SAFETY AND TOLERABILITY ANALYSIS

Safety and tolerability assessments will include adverse events (AEs), vital signs, and pulmonary function tests. If there is a difference between the ITT set and SAF set, then all safety summaries (or analyses if applicable) will be conducted using the SAF set. Otherwise, the ITT set will be used. No formal hypothesis testing will be performed to compare differences between treatment groups.

## 7.1 Extent of Exposure and Compliance

The number of doses received will be summarized by treatment group. The duration of study drug administration in minutes, the reason for study drug discontinuation, and whether 100% of study drug (4 mL) was delivered will be summarized for each dose by treatment group.




#### 7.2 Adverse Events

The AE reporting period for this study is continuous and begins at the time of randomization to study treatment and ends on Day 29. All AEs (both serious and nonserious) must be followed until resolution or until a stable clinical endpoint is reached. All measures required for AE management and the ultimate outcome of the AE must be recorded in the source documentation and in the eCRF.

AEs will be classified by SOC and PT using the most recent version of MedDRA.

# 7.2.1 Treatment-emergent Adverse Events

Treatment-emergent AEs are defined as those that begin or worsen after the start of study drug administration.

For adverse events with incomplete start dates, the same imputation algorithm for partial date information as described in Section 5.6 will be used for the determination of an AE being treatment emergent or not. Briefly, the unknown portions of an AE onset date will be imputed to the latest possible before being compared to the date of first study drug administration.

# 7.2.2 Adverse Event Severity

The severity (i.e., grade) of an AE will be assessed by the Investigator according to the definitions in the Common Terminology Criteria for Adverse Events (CTCAE) v5.0. If the AE is not specifically listed in the reference above, the following grades should be used:

- Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated
- Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting ageappropriate instrumental Activities of Daily Living (ADL)
- Grade 3 Severe or medically significant but not immediately life threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL
- Grade 4 Life-threatening consequences; urgent intervention indicated
- Grade 5 Death related to AE

## 7.2.3 Adverse Event Relationship to Study Drug

The Investigator must record his/her opinion concerning the relationship of the AE to study therapy (Unrelated, Unlikely, Possibly, Probably, Definitely) on the AE eCRF. See study protocol, Section 12.5 for details.

#### 7.2.4 Serious Adverse Events

An AE or suspected adverse reaction is considered "serious" if in the view of either the investigator or sponsor, it results in any of the following outcomes:

- Death
- A life-threatening adverse event
- In-patient hospitalization or prolongation of existing hospitalization




- Persistent or significant incapacity or substantial disruption to conduct normal life functions
- A congenital anomaly/birth defect
- Intervention to prevent any one of the other outcomes listed above (based on medical judgment)

#### 7.2.5 Adverse Event Summaries

All AEs (serious and non-serious) occurring after randomization and before the end of study, regardless of relationship to study drug, will be included and classified by SOC and PT using MedDRA.

For TEAEs, the following will be summarized and presented:

- i. An overall summary of TEAEs, which includes:
  - a. the number and percentage of subjects experiencing a TEAE
  - b. the number and percentage of subjects experiencing a TEAE by strongest relationship to study drug
  - c. the number and percentage of subjects experiencing a TEAE by greatest severity
  - d. the number and percentage of subjects experiencing a treatment-emergent SAE
  - e. the number and percentage of subjects experiencing a TEAE leading to death
  - f. the number and percentage of subjects experiencing a TEAE leading to study withdrawal
- ii. the number and percentage of subjects experiencing a TEAE by SOC and PT.
- iii. the number and percentage of subjects experiencing a potentially related TEAE by SOC and PT, where a potentially related TEAE is defined as any TEAE with a causal relationship to study drug assessed as 'Possibly Related', 'Probably Related', or 'Definitely Related'.
- iv. the number and percentage of subjects experiencing a TEAE by SOC, PT and the strongest relationship to study drug
- v. the number and percentage of subjects experiencing a TEAE by SOC, PT and the greatest severity
- vi. the number and percentage of subjects experiencing a treatment-emergent SAE by SOC and PT
- vii. the number and percentage of patients experiencing a TEAE leading to death by SOC and PT
- viii. the number and percentage of subjects experiencing a TEAE leading to study withdrawal by SOC and PT

In the overall summary of TEAEs table (i), besides tabulating the number and percentage of subjects, the total number of TEAE episodes will also be provided. If a subject has repeated episodes of a particular TEAE, all episodes will be counted in the summary table.




In the remaining summary tables, the incidence of TEAEs will be calculated by dividing the number of subjects who have experienced the event by the total number of subjects. Thus, the incidence of TEAEs is shown in terms of the total number of subjects and not in terms of the total number of episodes. If a subject has repeated episodes of a particular TEAE, only the most severe episode, or the episode with the strongest causal relationship to study drug, will be counted in the summary tables.

A subject with more than one type of TEAE in a particular SOC or PT will be counted only once in the total of subjects experiencing TEAEs in that particular SOC or PT.

All occurrences of all AEs and SAEs will be listed for each subject, grouped by treatment group. The listing will contain the following information: treatment group, verbatim term, SOC, PT, severity and grade (1-Mild, 2-Moderate, 3-Severe, 4-Life threatening, 5-Death), relationship to study drug, date and day of onset, date and day of resolution or death, action taken with regard to study drug, the outcome, whether the event was an SAE, whether it led to study withdrawal, and whether it is a TEAE. Listings will be sorted by treatment group, subject identification number, onset date, SOC, and PT. If the onset date is completely missing, then these events will be presented first. If the onset date is missing a month or a day, then these events will be presented before any complete dates.

# 7.3 Pulmonary Function Testing

Spirometry tests including FEV1 (L), % predicted FEV1, FVC (L), % predicted FVC and FEV1/FVC values will be collected at screening and FEV1 (L) will also be recorded at the time points presented in the Appendix A. FEV1 results will be summarized by presenting descriptive statistics of raw data of FEV1 (L) and percent change from each Pre-dose value to Post-dose value on the dosing days.

The proportion of subjects with percent decrease in FEV1 (L) from Pre-dose value to Post-dose value will be presented for each category: >10% and <=12% of reduction; >12% and <=20% of reduction; and >20% of reduction at each measurement time point (Day 1, Day 3, Day 6 and Day 10).

The percent change in FEV1 (L) from Pre-dose value to the protocol defined 30-min Post-dose values will be illustrated in a box/whisker graph on each dosing day by treatment group.

Spirometry results from unscheduled visits will be excluded from table summaries but will be included in the data listing.

# 7.4 Vital Signs

Descriptive summaries of pre and post treatment vital signs including systolic and diastolic blood pressure, pulse, respiratory rate, and body temperature will be prepared for each treatment group by visit.

A listing of all vital sign assessments throughout the study will be provided.

# 7.5 Other Safety Measures

Pregnancy test results, if applicable, will be presented in a listing.




#### 8. INTERIM ANALYSES

An external DSMB will be used to evaluate safety of the study in an ongoing manner. A full description of the membership, role, and responsibilities of the DSMB is provided in the DSMB charter. As specified there, a formal review of data will take place at DSMB meetings scheduled to occur after 40, 80 and 120 subjects have completed dosing.

As a further effort to ensure the safety of PUL-042, a stopping rule that is based only on mortality will be employed. A recommendation to stop the study would be made only if there is a high probability of excess mortality risk among subjects randomized to PUL-042. The following hierarchical analysis of mortality will be performed after 50% of subjects have been enrolled (50/group) and followed up for 28 days from the start of investigational therapy:

1) Based on blinded data, if no more than 3 deaths have occurred during the study this analysis will not be conducted due to the lack of evidence of increased mortality risk attributable to PUL-042.

#### If more than 3 deaths occur:

- 2) The Unblinded statistician will evaluate unblinded mortality data to determine the treatment specific death rate (i.e.,  $D_{Tx} = Deaths_{Tx} / N_{Tx}$ ; Tx = Active or Placebo).
- 3) If the difference,  $\Delta$ , in treatment-specific death rates (i.e.,  $\Delta = D_{Active} D_{Placebo}$ ) is greater than 7.5%, the DSMB will further review the totality of evidence and render a recommendation to the sponsor regarding study continuation.

#### Characteristics of this rule are as follows:

Assuming that the true underlying control arm mortality rate is 5% and using a normal approximation when comparing proportions, the probability of stopping is approximately:

- 90% if the true underlying mortality rate attributable to PUL-042 is 25%.
- 62% if the true underlying mortality rate attributable to PUL-042 is 15%.
- only 11% if the true underlying mortality rate attributable to PUL-042 is 5% (equal to the assumed true underlying control arm mortality rate).

#### 9. SAMPLE SIZE AND POWER CALCULATIONS

The trial size of 200 subjects (100 PUL-042 inhalation solution: 100 placebo) was chosen based on clinical considerations. The rates of infection to adequately estimate a sample size for a statistically significant result are unknown.

Enrolled subjects will be randomized with equal probability to receive blinded treatment consisting of either PUL-042 or placebo.

#### 10. REFERENCES

1. World Health Organization. WHO-COVID-19: Treatment Trial Design Master Protocol Synopsis, Draft February 18, 2020




#### 11. APPENDIX

# 11.1 Appendix A: Schedule of Events

| Event | Screening | Dose 1a | Dose 2, 3, 4 a | Follow-up/Early<br>Discontinuation from Study | Study Completion |
|---|---|---|---|---|---|
| | V1 | V2 | V3, 4, 5 | V6 | V7 |
| | Day -2 to Day 1 | Day 1b | Days 3, 6, 10 | Day 15 | Day 29 |
| Informed consent | X | | | | |
| Medical history | X | | | | |
| Pregnancy test <sup>c</sup> | X | | | X | X |
| Physical exam | X | X | X | X | |
| Vital signs <sup>d</sup> | X | X | X | X | |
| Spirometry <sup>e</sup> | X | X | X | | |
| Symptom score <sup>f</sup> | X | X | X | X | X |
| SARS-CoV-2 test <sup>g</sup> | | X | | X | X |
| Study drug administrationh | | X | X | | |
| Adverse events | X | X | X | X | X |
| Concomitant medications | X | X | X | X | X |
| Ordinal Scale for Clinical<br>Improvement | х | X | Х | X | Х |
| Randomization | X | | | | |

a Vital signs, adverse events, and concomitant medications will be assessed prior to administration of study medication and also at 30 minutes post-dose.


b There is no Day 0 in this study

<sup>&</sup>lt;sup>c</sup> Urine pregnancy test or serum pregnancy test if women are of child-bearing potential. If urine pregnancy test is positive, a serum pregnancy test must be done. Pregnancy test is required for Early Discontinuation, not Day 15.

d Vital signs will include body temperature, blood pressure measurements, heart rate, and respiratory rate.

Spirometry will be done at screening to document eligibility. On days of dosing, spirometry will be done pre-dose and at 30 minutes (±15) minutes post-dose. If the FEV1 is reduced > 10% compared to the pre-dose baseline the FEV1 should be repeated as clinically indicated

f SARS-CoV-2 symptoms will be assessed at each visit according to the Symptom Score

<sup>§</sup> SARS-CoV-2 testing will be performed pre-dose on Day 1 (Visit 2), Day 15 (Visit 6) and at Day 29 (Visit 7). Additional testing should be conducted at any point during the study when clinical symptoms are suggestive of potential COVID-19.

h Study drug administration must be done by a health care professional